CLINICAL TRIAL: NCT03204877
Title: Acute Metabolic Effects of Melatonin Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Mel06062017
Record Dates: First submitted 2017-06-06; First posted 2017-07-02 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Glucose Metabolism Disorders
Keywords: Melatonin; Insulin sensitivity; Insulin secretion; Incretin response
MeSH Terms: conditions — Glucose Metabolism Disorders; Insulin Resistance | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Active Comparator): Four capsules of Melatonin 10 mg is administered orally every hours for four hours during the study day.
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Four capsules of placebo is administered orally every hours for four hours during the study day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin — Oral capsules
  Arms: Melatonin
Other: Placebo — Oral capsules
  Arms: Placebo

SUMMARY:
Modern living is associated with an epidemic of type 2 diabetes mellitus (T2DM). Sleep disturbances are strong independent risk factors for incident diabetes. Melatonin has been implicated in regulation of circadian rhythm and sleep, but it is also ascribed anti-oxidative properties and effects on glucose homeostasis. A potential association between melatonin and T2DM has only been addressed in few human physiological studies, but the topic has received renewed interest since genetic-epidemiological studies have pointed to a role for melatonin in the development of the disease. In the current study, the investigators wish to examine whether treatment with synthetic melatonin induces physiological changes that affect the risk of developing type 2 diabetes. Two studies of the physiological effects of melatonin are included in the present protocol. In study A, the investigators will examine the acute effects of Melatonin on insulin secretion and insulin sensitivity using a Botnia clamp and in study B the investigators will examine the potential effects of Melatonin on the incretin response.

DETAILED DESCRIPTION:
Modern living is associated with an epidemic of type 2 diabetes mellitus (T2DM). Sleep disturbances such as insomnia and frequent awakenings are strong independent risk factors for incident diabetes with a magnitude of effect comparable to a family history of diabetes. Melatonin has been implicated in regulation of circadian rhythm and sleep, but it is also ascribed anti-oxidative properties and effects on glucose homeostasis. In pancreatic islets melatonin have dual effects depending on which signaling pathway is activated by receptor binding, thus both inhibitory and stimulatory effects on insulin secretion have been reported. The effect of melatonin on the secretion of gut hormones such as glucagon-like peptide 1 (GLP-1) and influence of melatonin on beta cell sensitivity to gut hormones is largely unknown, but the presence of the melatonin receptor in the gut suggests that it may have a role. A potential association between melatonin and T2DM has only been addressed in few human physiological studies, but the topic has received renewed interest since genetic-epidemiological studies have pointed to a role for melatonin in the development of the disease. Genetic mutations in the melatonin receptor which is predicted to change the physiological effects of melatonin have been found to increase the risk for T2DM. Additionally, low endogenous melatonin production has been linked to T2DM risk.

The aim of the present study is to examine whether treatment with synthetic melatonin induces physiological changes that affect the risk of developing type 2 diabetes.

Two studies of the physiological effects of melatonin are included in the present protocol:

Study A:

In order to study the acute effects of melatonin administration in healthy men, the investigators aim for assessing whether:

* Melatonin affects the substrate turn-over as evaluated by indirect calorimetry
* Melatonin has influence on the ability to secrete insulin as assessed by intravenous glucose tolerance test
* Melatonin affects the physiological effects of insulin as assessed by use of the hyperinsulinemic euglycemic clamp
* Genetic mutations in the melatonin receptor gene affect the treatment response to melatonin

Study B:

The investigators aim for examining if melatonin given to healthy men affects the secretion of the glucose-lowering gut hormone glucagon-like peptide 1 (GLP-1) and/or affect the glucose-lowering effects of GLP-1. Specifically, the aim is to assess whether:

* Melatonin affects the glucose excursions and insulin secretion during an oral glucose tolerance test
* Melatonin affects the secretion of GLP-1 during an oral glucose tolerance test
* Melatonin affects the incretin response as assessed by an isoglycemic glucose infusion

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 20-40 years
* BMI between 22-30 kg/m2
* Written consent prior to study participation

Exclusion Criteria:

* Diabetes or impaired glucose tolerance (fasting p-glucose ≥ 6.1mmol/L)
* Daily use of a prescription drug
* Shift work within the last year
* Travel across >2 time zones in the past three months
* Use of melatonin on a regular basis within the last year
* Severe illness
* High performance athletes
* Daily tobacco smoking
* Previous diagnosis of a sleep disorder
* Present or earlier alcohol or drug abuse
* Unable to give informed consent
* Allergy towards melatonin

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 2 hours (from t= 105 to 225 minutes)
  Insulin sensitivity is assessed by a hyperinsulinemic euglycemic clamp, unit: mg/kg/min
Insulin secretion | 1 hour (from t = 45 to 105 minutes)
  Insulin secretion is assessed by an intravenous glucose tolerance test, unit: pmol/L (insulin)
Incretin response | 4 hours (from t = 0 to 240 minutes)
  The incretin response is assessed by the difference in incretin hormones between an oral glucose tolerance test and an isoglycemic intravenous glucose infusion, unit: pmol/L (GIP, GLP-1)

SECONDARY OUTCOMES:
Inflammatory markers | Baseline t = -60 minutes and at t = 45 minutes
  Assessed by blood samples, unit: pg/mL
Substrate oxidation | From t=15 minutes to 45 minutes and from t=195 minutes to 225 minutes
  Substrate oxidation is assessed by indirect calorimetry. Glucose oxidation: unit: mg/kg/min; protein oxidation: unit: mg/kg/min; lipid oxidation: unit: mg/kg/min
Hormones | Baseline t = -60 minutes and at t = 45 minutes
  Hormones are assessed by blood samples. Units: C-peptide: pmol/L; Cortisol: ng/mL; Adiponectin: mg/L; IGF-I (ng/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedersen MGB, Lauritzen ES, Svart MV, Stoy J, Sondergaard E, Thomsen HH, Kampmann U, Bjerre M, Jessen N, Moller N, Rittig N. Nutrient sensing: LEAP2 concentration in response to fasting, glucose, lactate, and beta-hydroxybutyrate in healthy young males. Am J Clin Nutr. 2023 Dec;118(6):1091-1098. doi: 10.1016/j.ajcnut.2023.10.007. Epub 2023 Oct 14. PMID 37844838
- [Derived] Lauritzen ES, Stoy J, Baech-Laursen C, Grarup N, Jessen N, Hansen T, Moller N, Hartmann B, Holst JJ, Kampmann U. The Effect of Melatonin on Incretin Hormones: Results From Experimental and Randomized Clinical Studies. J Clin Endocrinol Metab. 2021 Nov 19;106(12):e5109-e5123. doi: 10.1210/clinem/dgab521. PMID 34265066
- [Derived] Kampmann U, Lauritzen ES, Grarup N, Jessen N, Hansen T, Moller N, Stoy J. Acute metabolic effects of melatonin-A randomized crossover study in healthy young men. J Pineal Res. 2021 Mar;70(2):e12706. doi: 10.1111/jpi.12706. Epub 2020 Dec 6. PMID 33220095